CLINICAL TRIAL: NCT05305326
Title: Telocytes in Placental Tissues of Patients With Gestational and Pre-gestational Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Othman Abdelkareem Mohammad Ahmad, Lecturer of Obstetrics and Gynecology, Sohag University
Other Study IDs: Soh-Med-21-12-39
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetes in Pregnancy
Keywords: pregnancy; diabetes; telocytes; placenta; umbilical cord
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fragments of the central part of the placenta Small section of the umbilical cord
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Singleton pregnancies undergoing elective pre-labour CS at gestational age (37+0 to 40+0) that are healthy
- Gestational diabetes: Singleton pregnancies complicated with gestational diabetes undergoing pre-labour CS at gestational age (37+0 to 40+0) that are otherwise healthy
- Type 1 diabetes with pregnancy: Singleton pregnancies complicated with Type 1 diabetes undergoing pre-labour CS at gestational age (37+0 to 40+0) that are otherwise healthy
- Type 2 diabetes with pregnancy: Singleton pregnancies complicated with Type 2 diabetes undergoing pre-labour CS at gestational age (37+0 to 40+0) that are otherwise healthy

SUMMARY:
Examining the expression of telocytes in the placental tissues and umbilical cord of patients with gestational or pregestational diabetes during pregnancy compared to control.

DETAILED DESCRIPTION:
this is an observational study, patients with gestational or pre-gestational diabetes undergoing elective (pre-labour) Cesarean section will be asked to participate in the study. Samples of placenta and umbilical cord will be taken postpartum and will be fixed and examined using immunohistochemistry to measure abundance of telocytes in these tissues. another group of patients with non complicated pregnancies will be asked to join as a control. As the topic was never studied before, a pilot phase of 10 patients per group will be done followed by sample size collection based on SD of number of telocytes in each group. Diabetes patients will divided in 3 subgroups; Gestational diabetes and pre-gestational diabetes type 1 or 2. Each group will be further subdivided according to HBA1C level collected at the time of delivery into controlled or non controlled.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women presented at the delivery ward in Sohag University Hospital, Sohag, Egypt with the following criteria:

  1. Study group: Singleton pregnancies complicated with diabetes undergoing pre-labour CS at gestational age (37+0 to 40+0). These will be divided into 3 groups according to the type of disease either Gestational diabetes (Group A), pregestational diabetes type 1 (Group B) or type 2 (Group C). 2-Control group: Singleton pregnancies undergoing elective pre-labour CS at gestational age (37+0 to 40+0) that are otherwise healthy

Exclusion Criteria:

* Women with history of medical co-morbidities other than diabetes are excluded from the study. This includes the following: Chronic hypertension, renal diseases, autoimmune diseases, history of organ transplantation and immunosuppressive therapy, hematological diseases, history of thrombotic events, cardiopulmonary diseases, liver diseases Acute and chronic inflammatory diseases.
* Pregnancy induced medical disorders like: Gestational hypertension, preeclampsia, Gestational thrombocytopenia, and proteinuria.
* Multiple pregnancies.
* Abnormal placentation, i.e. Placenta previa and Morbidly adherent placenta.
* Fetal anomalies.
* vaginal deliveries and CS in labor.
* Spontaneous delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women presented at the delivery ward in Sohag University Hospital, Sohag, Egypt fulfilling the inclusion criteria. A pilot phase will include 10 patients in each group. Based on primary analysis, proper sample size will be calculated.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Telocytes | Telocytes will be assessed in placental and umbilical cord tissues fixed immediately after delivery.
  number of telocytes per high power field detected by IHC

CONTACTS AND LOCATIONS:
Overall Officials: Amr O Abdelkareem, MD, Principal Investigator — Sohag Faculty of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
on personal request de-identified IPD could be shared in the form of Telocytes score of placenta and cord and statistical analysis done.
Supporting Information: Study Protocol
Time Frame: January 2024 and up to 5 years duration
Access Criteria: email amr.oth@med.sohag.edu.eg

REFERENCES:
- [Background] Blanco MV, Vega HR, Giuliano R, Grana DR, Azzato F, Lerman J, Milei J. Histomorphometry of umbilical cord blood vessels in preeclampsia. J Clin Hypertens (Greenwich). 2011 Jan;13(1):30-4. doi: 10.1111/j.1751-7176.2010.00384.x. Epub 2010 Nov 4. PMID 21214719
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Feig DS, Berger H, Donovan L, Godbout A, Kader T, Keely E, Sanghera R. Diabetes and Pregnancy. Can J Diabetes. 2018 Apr;42 Suppl 1:S255-S282. doi: 10.1016/j.jcjd.2017.10.038. No abstract available. PMID 29650105
- [Background] Feig DS, Razzaq A, Sykora K, Hux JE, Anderson GM. Trends in deliveries, prenatal care, and obstetrical complications in women with pregestational diabetes: a population-based study in Ontario, Canada, 1996-2001. Diabetes Care. 2006 Feb;29(2):232-5. doi: 10.2337/diacare.29.02.06.dc05-1482. PMID 16443865
- [Background] Nizyaeva NV, Sukhacheva TV, Serov RA, Kulikova GV, Nagovitsyna MN, Kan NE, Tyutyunnik VL, Pavlovich SV, Poltavtseva RA, Yarotskaya EL, Shchegolev AI, Sukhikh GT. Ultrastructural and Immunohistochemical Features of Telocytes in Placental Villi in Preeclampsia. Sci Rep. 2018 Feb 22;8(1):3453. doi: 10.1038/s41598-018-21492-w. PMID 29472628
- [Background] Chamberlain JJ, Rhinehart AS, Shaefer CF Jr, Neuman A. Diagnosis and Management of Diabetes: Synopsis of the 2016 American Diabetes Association Standards of Medical Care in Diabetes. Ann Intern Med. 2016 Apr 19;164(8):542-52. doi: 10.7326/M15-3016. Epub 2016 Mar 1. PMID 26928912
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693